CLINICAL TRIAL: NCT00863850
Title: Open-Label Study to Investigate the Pharmacokinetics of Bendamustine Hydrochloride Following Intravenous Infusion of [14C] Bendamustine Hydrochloride in Patients With Relapsed or Refractory Malignancy
Brief Title: Pharmacokinetics of Bendamustine Hydrochloride in Patients With Relapsed or Refractory Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C18083/1039/PK/NL
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Malignancy
MeSH Terms: conditions — Neoplasms | interventions — Bendamustine Hydrochloride

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bendamustine

INTERVENTIONS:
Drug: bendamustine — Bendamustine 120 mg/m2 on Days 1 and 2 every 28 days (one cycle) for up to 6 cycles. Radiolabeled [14C] bendamustine will be given on day 1 of cycle 1 only.

SUMMARY:
An Open-Label Study to Investigate the Pharmacokinetics of Bendamustine Hydrochloride in Patients With Relapsed or Refractory Malignancy (Hematologic or Nonhematologic)

ELIGIBILITY:
Key Inclusion Criteria:

* The patient must have a histologically or cytologically confirmed, relapsed or refractory malignancy, except for uveal melanoma, sarcoma or primary brain tumors. Additionally, the malignancy must be considered unresponsive or poorly responsive to accepted treatment modalities.
* The patient has a World Health Organization (WHO) performance status of 0-2.
* The patient has an estimated life expectancy of at least 3 months.
* The patient, if a woman, is surgically sterile, 2 years postmenopausal, or, if of child bearing potential, using a medically accepted method of contraception, and agrees to continued use of this method for the duration of the study and for 90 days after discontinuation of study drug. Acceptable methods of contraception include abstinence or an intrauterine device (IUD) known to have a failure rate of less than 1% per year.
* The patient, if a man, is surgically sterile, or, if capable of producing offspring, is currently using an approved method of birth control and agrees to continued use of this method for the duration of the study (and for 90 days after taking the last dose of study medication).
* Absolute neutrophil count (ANC) ≥1000 cells/mm3, platelet count ≥100000 cells/mm3, and hemoglobin greater than or equal to 9 g/dL.
* The patient has adequate hepatic function. For patients without liver metastases, adequate hepatic function is defined as ≤2.5 x upper limit of the normal range [ULN] for aspartate aminotransferase [AST] and alanine aminotransferase [ALT], and ≤1.5 x ULN for total bilirubin. For patients with liver metastases, adequate hepatic function is defined as ≤5 x ULN for AST and ALT, and ≤1.5 x ULN for total bilirubin. Patients with non-clinically significant elevations of bilirubin due to known or suspected Gilbert's disease are eligible; this must be documented on the medical history page of the case report form (CRF).
* The patient has a calculated creatinine clearance of >30 mL/minute as determined by the Cockcroft-Gault equation.

Key Exclusion Criteria:

* The patient has had chemotherapy, radiotherapy, radioimmunotherapy, or immunotherapy within 28 days prior to the first dose of study drug or has not recovered from adverse events due to any agents administered previously. For patients who received therapy with mitomycin C, the interval is 42 days.
* The patient has known cerebral metastases.
* The patient is receiving treatment other than bendamustine for hematologic/nonhematologic malignancy.
* The patient has had any previous treatment with bendamustine.
* The patient has been treated with any hematopoietic growth factors within 14 days of study entry (patients on chronic erythropoiesis stimulating agents are allowed).
* The patient is pregnant or lactating.
* The patient has had a serious infection, medical condition, or psychiatric condition that, in the opinion of the investigator, should preclude the patient from participating in the study.
* The patient has a known positive test result for human immunodeficiency virus (HIV) or a history of HIV disease.
* The patient has presence of inflammatory bowel disease, occlusion of the gastrointestinal tract, significant constipation, or any condition resulting in clinically significant obstruction of the urinary tract.
* The patient requires treatment with cytochrome P450 1A2 (CYP1A2) inducers or inhibitors on days 1 through 8 of cycle 1, has used CYP1A2 inhibitors within 14 days before the 1st administration of study drug, or has used CYP1A2 inducers within 30 days before the 1st administration of study drug.
* The patient is a smoker or an ex-smoker who stopped smoking less than 3 months before the 1st dose of study drug or is using or has used topical or oral nicotine preparations for smoking cessation within the past 3 months before the 1st dose of study drug.
* The patient has known hypersensitivity to bendamustine or any if its components (i.e., mannitol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Quantitative determination of the pharmacokinetics (distribution, metabolism, and excretion) of [14C]bendamustine and its metabolites in patients with confirmed, relapsed or refractory malignancy. | 168 hours (7 days)

SECONDARY OUTCOMES:
Safety and tolerability of bendamustine will be assessed throughout the study. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert - Sr. Director, Clinical Pharmacology, Study Director — Cephalon
Locations (1):
- Please Call For Information, Amsterdam, Netherlands